CLINICAL TRIAL: NCT06103318
Title: Cognitive Rehabilitation and Psychosocial Intervention Through a Stepped Digital Ecosystem in Breast Cancer: A Randomized Clinical Trial.
Brief Title: eHealth Interventions for Breast Cancer Cognitive Impairment
Acronym: ICOgnition
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Català d'Oncologia (Other)
Collaborators: Institut d'Investigació Biomèdica de Bellvitge (Other); Carlos III Health Institute (Other Government)
Responsible Party: Principal Investigator, Cristian Ochoa Arnedo, PhD, Clinical Psychologist, Institut Català d'Oncologia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI22/01255; PR270/22 (Other: Research Ethics Committee of Bellvitge University Hospital)
Record Dates: First submitted 2023-10-23; First posted 2023-10-26 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer; Cognitive Dysfunction
Keywords: eHealth; Breast Cancer; Cancer Related Cognitive Impairment (CRCI); Chemobrain; Psychoeducation; Cognitive Training; Emotional distress; Randomised Control Trial; Psycho-oncology; Digital Health; Quality of Life
MeSH Terms: conditions — Breast Neoplasms; Cognitive Dysfunction; Chemotherapy-Related Cognitive Impairment | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: The study proposes a superiority RCT with two parallel groups (online psychosocial care vs. online integrated and stepped cognitive intervention) with 1:1 allocation. The study design will contain 2 (treatment conditions) × 3 (follow-up assessments) factors.
Who Masked: Outcomes Assessor
Masking Description: To implement masking in the outcome assessor, the study will use an external service, the Biostatistical Services of The Bellvitge Biomedical Research Institute (IDIBELL). This external service will collect information through online questionnaires using REDCap, a secure web platform. Using an external service will help maintain the integrity of the study and prevents potential biases. Blinding in this context ensures that the assessment of outcomes is conducted impartially and without any influence from knowledge about the treatment assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICOnnectat (Active Comparator): ICOnnecta't is a stepped-care digital intervention tailored to breast cancer patients' psychosocial needs. It consists of four levels:
  1. rst level. Psychosocial Screening and Monitoring: Patients assess their emotional distress and symptoms; consultations with a health psychologist are scheduled if distress is high.
  2. nd level. Campus (Psychoeducation and Health Education): Patients access educational resources covering medical information, emotional well-being, relationships, and healthy habits.
  3. r level. Community Psychosocial Support: Patients engage in an online community to share experiences and concerns under supervision.
  4. th level. Online Group Psychotherapy: Patients participate in online group psychotherapy sessions led by a psycho-oncology specialist.
  Interventions: Behavioral: ICOgnition
- ICOgnition (Experimental): ICOgnition enhances ICOnnecta't with a Cognitive Module, following the same stepped-structure and specifically addressing cognitive deficits in breast cancer patients. It includes:
  1. rst level. Cognitive Screening and Monitoring: Patients complete monthly cognitive assessments and online objective cognitive tests. If scores indicate impairment, they advance to the next level.
  2. nd level. Cognitive Psychoeducational Campus: Patients undergo psychoeducation focusing on cognitive impairment understanding, behavioural strategies to enhance cognitive functioning, and acceptance strategies through mindfulness and metaphors.
  3. rd level. Online Cognitive Training: Individual 30-minute online cognitive training sessions are conducted twice a week for 12 weeks, targeting specific cognitive skills. Sessions are facilitated through the CogniFit program, integrated with the ICOnnecta't App.
  Interventions: Behavioral: ICOgnition

INTERVENTIONS:
Behavioral: ICOgnition — The ICOgnition intervention for breast cancer patients consists of three levels:
  Level 1: Monthly assessments using FACT-Cog PCI and Cognifit. Scores <54 (PCI) or ≤250 (Cognifit) escalate to Level 2.
  Level 2: Specialized content includes Cognitive Psychoeducation, validating experiences and improving health literacy; Behavioral Guidance, offering practical strategies for daily tasks; and Embracing Cognitive Deficits, promoting self-compassion and acceptance through mindfulness and metaphors.
  Level 3: Online cognitive training focuses on enhancing cognitive skills through gaming exercises, completing the comprehensive intervention approach.
  Other Names: Psychoeducational and Cognitive Training

SUMMARY:
This study investigates the effectiveness of integrating a cognitive rehabilitation module into a digital psychosocial intervention for recently diagnosed breast cancer patients. The trial involves 176 participants, with one group receiving the ICOnnecta't program (stepped psychosocial intervention) and the other receiving ICOnnecta't with an additional cognitive stepped intervention called ICOgnition. ICOgnition has three levels of intervention including cognitive screening and monitoring, psychoeducation, and online cognitive training. Assessments of the study outcomes will be conducted at baseline, 3 months, 6 months, and 1 year, measuring cognitive functioning, emotional well-being, medication adherence, work functioning, and overall quality of life. The study aims to improve understanding of efficient ways to detect cognitive dysfunction in cancer patients and assess the benefits and feasibility of this early intervention for managing cognitive impairment in breast cancer patients.

DETAILED DESCRIPTION:
BACKGROUND

Breast cancer (BC) diagnoses have increased, and while survival rates have improved, the focus on the quality of life (QoL) for survivors, including cognitive function, has intensified. Cancer-related cognitive impairment (CRCI) is recognized, encompassing objective deficits and subjective experiences. Various factors, such as chemotherapy agents, stress, and psychological factors, influence CRCI. Non-pharmacological treatments, including psychoeducational interventions and cognitive training, have shown promise. However, there are barriers in oncological settings, including a lack of awareness and standardized protocols. Current developed technologies like eHealth offer solutions, yet studies addressing cognitive care in eHealth psychosocial interventions are limited. This study aims to assess the ICOgnition digital intervention's effectiveness in improving BC patients' subjective and objective cognitive symptoms. It also explores factors influencing cognitive function, the effectiveness of online cognitive testing, and the gap between objective and subjective deficits. The study will also evaluate the feasibility and cost-effectiveness of ICOnnecta't + ICOgnition interventions to provide insights into their scalability and sustainability. The hypothesis suggests that the ICOnnecta't-enhanced intervention (ICOgnition) will outperform ICOnnecta't alone in improving both subjective and objective cognitive functioning in BC patients.

METHODS/DESIGN

The trial is conducted at the Catalan Institute of Oncology (ICO) in Hospitalet de Llobregat. Patients meeting inclusion criteria are referred by the Breast Functional Unit to the ICOnnecta't Program team. Eligible candidates receive detailed study information via a call and, if willing to participate, schedule an in-person appointment at the ICOnnecta't Space. Researchers explain the study, obtain informed consent, and utilize the secure web platform REDCap for questionnaires. Assessments occur at baseline (T1), 3 months (T2), 6 months (T3), and 12 months (T4). Recruitment starts in December 2023 and spans a year.

Breast cancer patients will be randomly assigned to one of the two treatment groups using REDCap, employing a simple randomization method (1:1).

o Study Sample

The study will include 176 female breast cancer patients in the acute survival phase from ICO Hospitalet.

o Statistical Analysis:

Primary Outcome Analysis

The study will employ independent Linear Mixed Models with patients clustered to analyze cognitive outcomes between the two intervention groups: digital stepped psychosocial care vs. digital stepped psychosocial care + cognitive module. Subjective Cognition (FACT-Cog) and Objective Cognition (Neurocognitive Index) will be separately assessed, adjusting for age and education. Descriptive statistics, effect sizes, and 95% confidence intervals will be reported.

Secondary Outcome Analysis

Linear Mixed Models will be used to analyze secondary outcomes (e.g., depression, anxiety, distress, quality of life) following the same procedure. Mediation analysis will explore emotional distress and posttraumatic stress as mediators between interventions and cognitive responses.

Other Pre-Specified Outcome Analyses

* Discrepancy between Objective and Subjective Measures: Standardized values will be compared using ICC, Bland-Altman Plot, and linear regression to identify variables explaining discrepancies.
* Clusters of Cognitive Impairment: Cluster analysis will identify participant groups with similar cognitive profiles and explore differences in demographics, clinical variables, and treatment response.
* Cognitive Assessment Optimization: The equivalence of online vs. paper and pencil tests in detecting cognitive impairment will be tested, and the most sensitive test for CRCI detection will be explored.
* Cost-Utility Analysis: This analysis expresses the cost-effectiveness of interventions in terms of cost per Quality-Adjusted Life Year (QALY) gained, a common measure used in healthcare decision-making.

  * Statistical Power:

Utilizing GLIPMPSE, the study has a power of 0.802 with a significance level of 0.05. With 176 subjects (88 in each group), the study can detect a significant difference of 5.9 units, assuming a common standard deviation of 15, based on previous research findings (Bell et al., 2018).

o Discussion

The ICOgnition intervention offers a promising and comprehensive approach to address cognitive difficulties in newly diagnosed breast cancer patients. By integrating digital psychosocial support, personalized cognitive training, and psychoeducational resources, this intervention aims to enhance cognitive function and improve the overall quality of life for patients. Notably, its potential impact could extend to individuals facing cognitive challenges in various medical conditions beyond breast cancer. However, challenges related to implementation, resource allocation, patient adherence, and economic evaluation need careful consideration to ensure the intervention's effectiveness in real-world settings. If successfully implemented, ICOgnition could serve as a valuable model for addressing cognitive impairments, fostering a better understanding of cognitive challenges in medical settings, and enhancing patients' overall well-being.

ELIGIBILITY:
Inclusion Criteria:

* Women within 6 weeks after a Breast Cancer diagnosis
* Having online access and a user-level knowledge of the internet
* Understanding of Spanish language

Exclusion Criteria:

* Any additional medical condition that may affect neuropsychological performance
* Presence of a psychiatric condition including substance use disorders in the last 3 months (excluding tobacco addiction)
* Significant autolytic ideation

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2024-03-14 (Estimated); Primary Completion 2025-04-07 (Estimated); Study Completion 2025-09-07 (Estimated)

PRIMARY OUTCOMES:
Change in Subjective cognition | Assessment will be conducted at baseline and at 3 months, 6 months and 12 months
  The Functional Assessment of Cancer Therapy-Cognitive Function, FACT-Cog, Perceived Cognitive Impairment sub-scale (PCI), developed specifically to assess cognitive difficulties in cancer patients (https://www.facit.org/measures/FACT-Cog) is used. Lower scores (0-72) indicate a poor perceived performance.
Change in Objective Cognition (Digital assessment) | Assessment will be conducted at baseline and at 12 months
  The objective cognitive assessment will be provided by the licensed computer program CogniFit Inc © 2023. CogniFit offers a specific cognitive assessment called "Chemfog," which measures 6 cognitive domains: planning, processing speed, short-term memory, focus attention, coordination and spatial perception. Lower scores (0-800) indicate poor objective performance in those domains.
Change in Objective Cognition (Paper and pencil assessment) | Assessment will be conducted at baseline and at 12 months
  Verbal Learning, Immediate Verbal Memory and Delayed Verbal Memory will be measured through RAVLT - Rey Auditory Verbal Learning Test. The executive functions domains that will be measured are cognitive flexibility through Trail Making Test B (TMT-B) [50], verbal fluency through its Spanish version and working memory through Digit Span backward of the Wechsler Adult Intelligence Scale IV (WAIS-IV). Attention will be measured via TMT-A and Digit Span forward (WAIS-IV). Finally, Digit Symbol Substitution Test (DSST; WAIS-IV) will be used to measure processing speed.

SECONDARY OUTCOMES:
Change in emotional distress | Assessment will be conducted at baseline and at 3 months, 6 months and 12 months
  Hospital Anxiety and Depression Scale (HADS) will be used to assess emotional distress through 7 anxiety items (HADS-Anxiety) and 7 depression items (HADS-Depression). The range of scores is 0-21 for each subscale, and 0-42 for the overall questionnaire, where higher scores indicate worse clinical symptoms
Change in Medication adherence | Assessment will be conducted at baseline and at 3 months, 6 months and 12 months
  Medication adherence will be assessed through the Spanish version of Adherence to Refill and Medication Scale (ARMS-e), which is a valid and reliable scale for patients with chronic disease. This instrument consists of 12 questions: 8 are focused on the patient's consistency in taking medication appropriately and 4 on their proper collection. Lower overall scores correspond to better adherence.
Change in Quality of Life | Assessment will be conducted at baseline and at 12 months
  The European Quality of Life Scale (EQ-5D- 3L) provides a measure of Health-Related QoL (HRQoL) and is helpful for the evaluation of the cost-utility of health interventions. Lower scores represent worst health status.
Post-traumatic Stress | Assessment will be conducted at baseline and at 12 months
  The Post-traumatic Stress Disorder Checklist (PCL-5) is widely used in clinical and research settings to screen for post-traumatic symptoms. Higher scores indicate a higher severity of post-traumatic symptoms
Changes in Work role functioning | Assessment will be conducted at baseline and at 12 months
  Work Role Functioning Questionnaire (WRFQ): a self-report assessment tool, validated in cancer patients and in Spanish population, that is used to evaluate an individual's work-related functioning and productivity. It is specifically designed to measure how mental health symptoms and conditions impact an individual's ability to perform in a work environment. Higher scores indicate better work-related functioning.
Changes in Health Literacy | Assessment will be conducted at baseline and at 12 months
  Health literacy will be measured with a visual analogue scale with the following question (translated from Spanish): "Please indicate your level of satisfaction with the information provided to you by the Catalan Institute of Oncology (ICO) regarding your illness and treatments, where 0 is very dissatisfied with the information received, and 10 is very satisfied with the information received ".
Intervention Satisfaction | Assessment will be conducted at 3 months
  Intervention Satisfaction will be measured with a visual analogue scale with the following question (translated from Spanish): "Rate from 0 to 10 to what extent you are satisfied with the ICOnnecta't/ICognition Intervention, where 0 is completely dissatisfied and 10 is completely satisfied".
ICOnnecta't / ICOgnition App Usability | Assessment will be conducted at 3 months
  App Usability will be measured with a visual analogue scale with the following question (translated from Spanish): "Rate from 0 to 10 to what extent you found the application easy to use, where 0 is very difficult to use and 10 is very easy to use"

OTHER OUTCOMES:
Work absenteeism | 12 months post-intervention
  Number of days of patients' sick leaves (Electronic Health Record).
Professionals' salaries | 12 months post-intervention
  Number of professionals involved in the ICOnnecta't treatment or ICOnnecta't + ICOgnition platform as well as the number of professionals' working hours per week and costs (Electronic Health Record).
Infrastructure costs | 12 months post-intervention
  Costs per user and per month for the development and maintenance of the ICOnnecta't + ICOgnition platform (experimental group) and costs of ICOnnecta't platform alone per user and month.
Psychotropic Medication | 12 months post-intervention
  First, the Electronic Health Record will be checked to collect psychotropic medication data for each group during the study. Second, the pharmacy service of ICO will calculate the medication costs.

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Ochoa Arnedo, PhD, Principal Investigator — Institut Català d'Oncologia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Farrell E, Smith A, Collins B. Objective-subjective disparity in cancer-related cognitive impairment: does the use of change measures help reconcile the difference? Psychooncology. 2017 Oct;26(10):1667-1674. doi: 10.1002/pon.4190. Epub 2016 Jul 14. PMID 27278814
- [Background] Eide S, Feng ZP. Doxorubicin chemotherapy-induced "chemo-brain": Meta-analysis. Eur J Pharmacol. 2020 Aug 15;881:173078. doi: 10.1016/j.ejphar.2020.173078. Epub 2020 Jun 5. PMID 32505665
- [Background] Jim HS, Phillips KM, Chait S, Faul LA, Popa MA, Lee YH, Hussin MG, Jacobsen PB, Small BJ. Meta-analysis of cognitive functioning in breast cancer survivors previously treated with standard-dose chemotherapy. J Clin Oncol. 2012 Oct 10;30(29):3578-87. doi: 10.1200/JCO.2011.39.5640. Epub 2012 Aug 27. PMID 22927526
- [Background] Stewart A, Bielajew C, Collins B, Parkinson M, Tomiak E. A meta-analysis of the neuropsychological effects of adjuvant chemotherapy treatment in women treated for breast cancer. Clin Neuropsychol. 2006 Feb;20(1):76-89. doi: 10.1080/138540491005875. PMID 16410227
- [Background] Lange M, Joly F, Vardy J, Ahles T, Dubois M, Tron L, Winocur G, De Ruiter MB, Castel H. Cancer-related cognitive impairment: an update on state of the art, detection, and management strategies in cancer survivors. Ann Oncol. 2019 Dec 1;30(12):1925-1940. doi: 10.1093/annonc/mdz410. PMID 31617564
- [Background] Boscher C, Joly F, Clarisse B, Humbert X, Grellard JM, Binarelli G, Tron L, Licaj I, Lange M. Perceived Cognitive Impairment in Breast Cancer Survivors and Its Relationships with Psychological Factors. Cancers (Basel). 2020 Oct 16;12(10):3000. doi: 10.3390/cancers12103000. PMID 33081111
- [Background] Mackenzie L, Marshall K. Effective non-pharmacological interventions for cancer related cognitive impairment in adults (excluding central nervous system or head and neck cancer): systematic review and meta-analysis. Eur J Phys Rehabil Med. 2022 Apr;58(2):258-270. doi: 10.23736/S1973-9087.21.06898-2. Epub 2021 Sep 9. PMID 34498828
- [Background] Treanor CJ, McMenamin UC, O'Neill RF, Cardwell CR, Clarke MJ, Cantwell M, Donnelly M. Non-pharmacological interventions for cognitive impairment due to systemic cancer treatment. Cochrane Database Syst Rev. 2016 Aug 16;2016(8):CD011325. doi: 10.1002/14651858.CD011325.pub2. PMID 27529826
- [Background] Kim Y, Kang SJ. Computerized programs for cancer survivors with cognitive problems: a systematic review. J Cancer Surviv. 2019 Dec;13(6):911-920. doi: 10.1007/s11764-019-00807-4. Epub 2019 Oct 5. PMID 31587187
- [Background] Binarelli G, Joly F, Tron L, Lefevre Arbogast S, Lange M. Management of Cancer-Related Cognitive Impairment: A Systematic Review of Computerized Cognitive Stimulation and Computerized Physical Activity. Cancers (Basel). 2021 Oct 14;13(20):5161. doi: 10.3390/cancers13205161. PMID 34680310
- [Background] Binarelli G, Lange M, Dos Santos M, Grellard JM, Lelaidier A, Tron L, Lefevre Arbogast S, Clarisse B, Joly F. Multimodal Web-Based Intervention for Cancer-Related Cognitive Impairment in Breast Cancer Patients: Cog-Stim Feasibility Study Protocol. Cancers (Basel). 2021 Sep 28;13(19):4868. doi: 10.3390/cancers13194868. PMID 34638354
- [Background] Penedo FJ, Oswald LB, Kronenfeld JP, Garcia SF, Cella D, Yanez B. The increasing value of eHealth in the delivery of patient-centred cancer care. Lancet Oncol. 2020 May;21(5):e240-e251. doi: 10.1016/S1470-2045(20)30021-8. PMID 32359500
- [Background] Medina JC, Flix-Valle A, Rodriguez-Ortega A, Hernandez-Ribas R, Lleras de Frutos M, Ochoa-Arnedo C. ICOnnecta't: Development and Initial Results of a Stepped Psychosocial eHealth Ecosystem to Facilitate Risk Assessment and Prevention of Early Emotional Distress in Breast Cancer Survivors' Journey. Cancers (Basel). 2022 Feb 15;14(4):974. doi: 10.3390/cancers14040974. PMID 35205722
- [Background] Kaiser J, Dietrich J, Amiri M, Ruschel I, Akbaba H, Hantke N, Fliessbach K, Senf B, Solbach C, Bledowski C. Cognitive Performance and Psychological Distress in Breast Cancer Patients at Disease Onset. Front Psychol. 2019 Nov 15;10:2584. doi: 10.3389/fpsyg.2019.02584. eCollection 2019. PMID 31803117
- [Background] Ciria-Suarez L, Costas L, Flix-Valle A, Serra-Blasco M, Medina JC, Ochoa-Arnedo C. A Digital Cancer Ecosystem to Deliver Health and Psychosocial Education as Preventive Intervention. Cancers (Basel). 2022 Jul 30;14(15):3724. doi: 10.3390/cancers14153724. PMID 35954388
- [Background] Fardell JE, Bray V, Bell ML, Rabe B, Dhillon H, Vardy JL. Screening for cognitive symptoms among cancer patients during chemotherapy: Sensitivity and specificity of a single item self-report cognitive change score. Psychooncology. 2022 Aug;31(8):1294-1301. doi: 10.1002/pon.5928. Epub 2022 Mar 30. PMID 35320617
- [Background] Bell ML, Dhillon HM, Bray VJ, Vardy JL. Important differences and meaningful changes for the functional assessment of cancer therapy-cognitive function (FACT-COG). J Patient-Reported Outcomes 2018;2:48.
- [Background] Shari NI, Zainal NZ, Ng CG. Effects of brief acceptance and commitment therapy (ACT) on subjective cognitive impairment in breast cancer patients undergoing chemotherapy. J Psychosoc Oncol. 2021;39(6):695-714. doi: 10.1080/07347332.2020.1856283. Epub 2020 Dec 8. PMID 33287685
- [Background] Henneghan AM, Van Dyk K, Kaufmann T, Harrison R, Gibbons C, Heijnen C, Kesler SR. Measuring Self-Reported Cancer-Related Cognitive Impairment: Recommendations From the Cancer Neuroscience Initiative Working Group. J Natl Cancer Inst. 2021 Nov 29;113(12):1625-1633. doi: 10.1093/jnci/djab027. PMID 33638633
- [Background] Kennedy-Martin M, Slaap B, Herdman M, van Reenen M, Kennedy-Martin T, Greiner W, Busschbach J, Boye KS. Which multi-attribute utility instruments are recommended for use in cost-utility analysis? A review of national health technology assessment (HTA) guidelines. Eur J Health Econ. 2020 Nov;21(8):1245-1257. doi: 10.1007/s10198-020-01195-8. Epub 2020 Jun 8. PMID 32514643
- [Derived] Serra-Blasco M, Souto-Sampera A, Medina JC, Flix-Valle A, Ciria-Suarez L, Arizu-Onassis A, Ruiz-Romeo M, Jansen F, Rodriguez A, Pernas S, Ochoa-Arnedo C. Cognitive-enhanced eHealth psychosocial stepped intervention for managing breast cancer-related cognitive impairment: Protocol for a randomized controlled trial. Digit Health. 2024 Jul 25;10:20552076241257082. doi: 10.1177/20552076241257082. eCollection 2024 Jan-Dec. PMID 39070895